CLINICAL TRIAL: NCT03144193
Title: Assessment of Efficacy in Daily Use of a Novel Skin Care Product (CG Skin Ltd.) for the Treatment of Photoaged Skin
Brief Title: Efficacy in Daily Use of a Novel Skin Care Product for the Treatment of Photoaged Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Rachel Watson, Reader in Dermatology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CGC03
Record Dates: First submitted 2017-03-27; First posted 2017-05-08 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Photoaging
Keywords: topical treatment; wrinkles; extracellular matrix

STUDY DESIGN:
Intervention Model Description: Assessment of efficacy of a novel anti-aging topical treatment compared to a placebo control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Topical anti-aging cosmetic cream (active)
  Interventions: Other: Topical anti-aging cosmetic cream
- Placebo (Placebo Comparator): Basic formulation without active ingredients (vehicle)
  Interventions: Other: Topical anti-aging cosmetic cream

INTERVENTIONS:
Other: Topical anti-aging cosmetic cream — Topical anti-aging cosmetic cream

SUMMARY:
Photoaged or chronically sun-exposed skin is characterised by a number of clinical features including fine and coarse wrinkles. The pathogenesis of wrinkle formation has yet to be determined fully but recent work suggests that ultraviolet radiation-induced reduction in dermal fibrillin (in the form of fibrillin-rich microfibrils) is important. Using an extended in vivo patch test assay, it has been identified that skin care products - currently marketed by CG Skin Ltd - increase the deposition of these microfibrils in photoaged dermis and hence have the potential to repair photoaged skin. The Investigators now propose to examine the efficacy of the product in randomized, placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Subjects who satisfy the inclusion/exclusion criteria and who have given their written, witnessed, informed consent will be admitted to the studies. Subjects will be clinically assessed (fine wrinkling, coarse wrinkling, mottled hyperpigmentation, sallowness) and clinical photographs taken prior to instruction on the use of the allocated cream by the study Investigator (product or placebo). Product will be applied daily to the entire face and dorsum of hands, including the wrists and extensor forearm, for six months. Successive follow-up visits (3 visits over a 6-month period) will be made to assess efficacy and safety. Subjects will be randomly allocated to self-treatment with either product or placebo cream using a computer generated code (Research Randomizer; www.randomizer.org).

The primary outcome measure will be treatment efficacy; this will be assessed by the study Investigators as changes in the clinical parameters of photoaging (fine wrinkles, coarse wrinkles, mottled hyperpigmentation, sallowness).

The Investigators will assess two secondary outcome measures: (1) Histological improvement in skin structure. Skin biopsies from the treated extensor forearm will be taken at study initiation and at the end of the six month study period. These biopsies will be evaluated for: (a) epidermal thickness; (b) fibrillin expression and; (c) pro-collagen I expression. (2) Tolerance and irritancy. Tolerance and irritation assessments will be made by recording the occurrence and severity of signs of erythema and scaling. Safety will be evaluated by recording all adverse events experienced by subjects. Any subject exhibiting adverse events of sufficient severity will be withdrawn from the trial. Completion or withdrawal of subjects from the trial will be noted on the end of study form. All subjects will be monitored for the occurrence of serious adverse events up to, and including, 28 days after their involvement with this study.

The trial will be conducted according to the recommendations of ICH GCP and those of the Declaration of Helsinki, only after approval of the study has been obtained from the relevant Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe photoaging of facial skin (grade 6 or above on the Griffiths scale);
* Willing to submit to examination of facial skin, hands and forearms;
* Willing to submit to self-treatment with product or placebo cream on face, hands and forearms, including wrists and extensor forearms, for 6 months;
* Willing to submit to clinical photography;
* Willing to submit to 3 mm punch biopsies from the wrist at beginning and end of trial;
* Signed informed consent.

Exclusion Criteria:

* Skin disease that would impair evaluation of the test sites;
* Topical or systemic retinoid within the past 6 months and 12 months respectively prior to entry to the study;
* Topical steroid or other topical drugs at treatment sites for at least two weeks prior to study entry;
* History of use of experimental drug or experimental device in the 30 days prior to entry into the study;
* Any significant cosmetic treatment for skin rejuvenation i.e. dermabrasion, chemical peels, face-lifts;
* Known allergy to any of the product or placebo ingredients;
* History of keloid scars.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinical appearance using a validated photonumeric wrinkle scale | Six (6) months
  Change in grade of facial wrinkles as assessed by a clinically competent researcher, using a validated photonumeric wrinkle scale (Griffiths et al., Arch Dermatol., 1992). Assessment of wrinkle grade will be made at baseline and at each follow-up appointment; clinical photography will be performed at each visit for subsequent quantitative image analysis of wrinkle effacement.

SECONDARY OUTCOMES:
Histological improvement in skin structure | Six (6) months
  Histology to assess dermal elastic fibres and the collagenous extracellular matrix
Tolerance and irritancy | Up to seven (7) months
  Assessments will be made by recording the occurrence and severity of signs of erythema and scaling

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E Watson, PhD, Principal Investigator — University of Manchester
Locations (1):
- Dermatopharmacology Unit, Salford Royal NHS Foundation Trust, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Source data will be shared with the study funder (CG Skin Ltd) on completion of the study and will collaborators at the University's Biostatistics Collaboration Unit.

REFERENCES:
- [Background] Watson RE, Griffiths CE, Craven NM, Shuttleworth CA, Kielty CM. Fibrillin-rich microfibrils are reduced in photoaged skin. Distribution at the dermal-epidermal junction. J Invest Dermatol. 1999 May;112(5):782-7. doi: 10.1046/j.1523-1747.1999.00562.x. PMID 10233772
- [Background] Watson RE, Craven NM, Kang S, Jones CJ, Kielty CM, Griffiths CE. A short-term screening protocol, using fibrillin-1 as a reporter molecule, for photoaging repair agents. J Invest Dermatol. 2001 May;116(5):672-8. doi: 10.1046/j.1523-1747.2001.01322.x. PMID 11348454
- [Background] Watson RE, Long SP, Bowden JJ, Bastrilles JY, Barton SP, Griffiths CE. Repair of photoaged dermal matrix by topical application of a cosmetic 'antiageing' product. Br J Dermatol. 2008 Mar;158(3):472-7. doi: 10.1111/j.1365-2133.2007.08364.x. Epub 2007 Dec 6. PMID 18070204
- [Background] Griffiths CE, Wang TS, Hamilton TA, Voorhees JJ, Ellis CN. A photonumeric scale for the assessment of cutaneous photodamage. Arch Dermatol. 1992 Mar;128(3):347-51. PMID 1550366